CLINICAL TRIAL: NCT00112255
Title: Partner Notification for Chlamydia in Primary Care: Randomised Controlled Trial and Economic Evaluation
Brief Title: Partner Notification for Chlamydia in Primary Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bristol (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HTA_97/32/31
Record Dates: First submitted 2005-05-31; First posted 2005-06-01 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Chlamydia Infections
Keywords: Chlamydia trachomatis; Chlamydia infections; Randomized controlled trials; Contact tracing; Family practice
MeSH Terms: conditions — Chlamydia Infections

INTERVENTIONS:
Behavioral: Practice nurse-led partner notification
Behavioral: Referral to specialist genitourinary clinic

SUMMARY:
The purpose of this study was to compare the effectiveness of partner notification by general practice nurses with referral to a specialist clinic for people with genital chlamydia diagnosed in a community setting. We hypothesised that referral to a specialist would be more effective in ensuring treatment of the sexual partners of infected people than the simpler nurse-led strategy.

DETAILED DESCRIPTION:
Partner notification (contact tracing) is essential to the control of sexually transmitted infections. Reports of new chlamydia infections have increased by 66% in the past five years. A National Chlamydia Screening Programme in England, and increasing primary care provision of sexual health care are part of the United Kingdom Government's strategy for tackling increasing rates of sexually transmitted infections. New strategies for managing chlamydia in non-specialist settings are urgently required: genitourinary medicine clinics are failing to cope with their increasing workload; and 45% of cases detected in the chlamydia screening pilot studies were diagnosed in general practice.

Partner notification involves informing the sexual partners of someone with a sexually transmitted infection of the possibility of exposure, offering them diagnosis and treatment, and providing advice about preventing future infection. In the United Kingdom, this is usually done by specialist sexual health advisers in departments of genitourinary medicine. The effectiveness of partner notification in non-specialist settings in developed countries is not known. We conducted a randomised controlled trial to compare the effectiveness of practice nurse-led partner notification with referral to a genitourinary clinic for partner notification conducted by a specialist health adviser, and to compare the resources used by each strategy.

Comparisons: Partner notification at the time of receiving diagnosis and treatment by general practice nurses who received a one-day training course and ongoing support by telephone calls or visits from a specialist adviser in sexual health, compared with referral to a genitourinary medicine clinic for partner notification by a specialist adviser in sexual health.

ELIGIBILITY:
Inclusion Criteria:

* Chlamydia trachomatis diagnosed through a population-based screening study
* Chlamydia test result received at patient's general practice
* Chlamydia cases diagnosed in general practice

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214
Dates: Start 2001-03; Study Completion 2002-12

PRIMARY OUTCOMES:
Percentage of index cases with at least one sexual partner treated
Number of sexual partners per index case treated

SECONDARY OUTCOMES:
Number of sexual partners per index case elicited during sexual history taking
Positive chlamydia test result six weeks after treatment
Adherence to advice to abstain from sexual intercourse until both partners completed treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Low, MFPH, Study Director — Chlamydia Screening Studies (ClaSS) Project General Practices
Locations (2):
- United Kingdom (2):
  - Chlamydia Screening Studies (ClaSS) project general practices, Bristol, Avon
  - Chlamydia Screening Studies (ClaSS) project general practices, Birmingham, West Midlands

REFERENCES:
- [Background] Low N, McCarthy A, Macleod J, Salisbury C, Horner PJ, Roberts TE, Campbell R, Herring A, Skidmore S, Sanford E, Sterne JA, Davey Smith G, Graham A, Huengsberg M, Ross J, Egger M. The chlamydia screening studies: rationale and design. Sex Transm Infect. 2004 Oct;80(5):342-8. doi: 10.1136/sti.2003.006197. PMID 15459400
- [Result] Low N, McCarthy A, Roberts TE, Huengsberg M, Sanford E, Sterne JA, Macleod J, Salisbury C, Pye K, Holloway A, Morcom A, Patel R, Robinson SM, Horner P, Barton PM, Egger M. Partner notification of chlamydia infection in primary care: randomised controlled trial and analysis of resource use. BMJ. 2006 Jan 7;332(7532):14-9. doi: 10.1136/bmj.38678.405370.7C. Epub 2005 Dec 15. PMID 16356945